CLINICAL TRIAL: NCT03900754
Title: A Pharmaco-imaging Approach to Predicting Social Functioning and Clinical Responses to Oxytocin Administration in Schizophrenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate Subject Recruitment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other); VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHBB-011-18F; 19-27265 (Other: University of California, San Francisco); 1I01CX001761-01A2 (NIH)
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Oxytocin
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: The study uses a combined within- and between-subject placebo-controlled study design. After screening, participants will be randomized into two study arms for the fMRI phase of the study. In each study arm, participants will complete a placebo-controlled, within-subject, pharmaco fMRI paradigm with one of two possible dosages of oxytocin (20 or 40IU) and placebo. 75 participants will be randomized to receive 20IU oxytocin and placebo and 75 will be randomized to receive 40IU oxytocin and placebo, with the order of administration randomized and separated by two weeks. Following the fMRI phase of the study, participants will be randomized to receive the same dosage of oxytocin the participant received in the fMRI phase, or placebo, twice daily for 3 weeks.
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal Oxytocin (Experimental): Dosages of oxytocin: 20IU or 40IU.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Intranasal administration of oxytocin
  Other Names: Syntocinon
  Arms: Intranasal Oxytocin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Schizophrenia has a devastating and disproportionate effect on veterans compared to the general US population. Some of the most disabling symptoms, such as low motivation, difficulty expressing emotions, and decreased ability to infer the mental states of others, cause poor social functioning. This means that veterans with schizophrenia have trouble navigating interpersonal interactions and building meaningful relationships in the community. Unfortunately, current antipsychotic medications typically only improve positive symptoms but fail to improve social functioning deficits, which are strong predictors of poor quality of life and functional outcomes. Oxytocin, a peptide found in the brain, plays an important role in social behavior and is known to moderate affiliation, stress, and learning across taxa. In this study, the investigators will test whether oxytocin could be an effective treatment for social functioning deficits in schizophrenia. The investigators will examine changes in brain activation to understand how oxytocin affects behavior and to predict which individuals may benefit from oxytocin treatment.

DETAILED DESCRIPTION:
The study uses a combined within- and between-subject placebo-controlled study design.

Within subjects phase: After screening, participants will be randomized into two study arms for the fMRI phase of the study. In each study arm, participants will complete a placebo-controlled, within-subject, pharmaco-fMRI paradigm with one of two possible dosages of oxytocin (20 or 40IU) and placebo. Following the fMRI phase of the study, participants will be randomized for the next phase of the study

Between subjects phase: Participants will receive the same dosage of oxytocin the participant received in the fMRI phase, or placebo, twice daily for 3 weeks. Before and after the three weeks of drug administration, participants will be assessed for social functioning, social ability, negative symptoms, and theory of mind. More participants will be randomized to receive chronically administered oxytocin than placebo to maximize the study's power to test the investigators' hypothesis that acute oxytocin-induced increases in right temporo-parietal junction activity will be positively correlated with improvements in social functioning (primary outcome), social ability, negative symptoms, and theory of mind over three weeks of oxytocin administration.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* age 18-70
* a diagnosis of schizophrenia, schizophreniform, schizoaffective, or brief psychotic disorder determined by the Structured Clinical Interview for DSM-5
* no medication changes or psychiatric hospitalizations in the past month
* SFS modified raw score of no more than 75

Exclusion Criteria:

* substance use disorder in the past month, except mild to moderate cannabis use disorder
* illness affecting the nasal passages
* significant neurological/medical disorder
* pacemakers
* extensive dental work
* claustrophobia
* deafness
* inability to read
* currently participating in a psychosocial intervention targeting social functioning deficits
* currently taking high dose testosterone or estrogen/progesterone
* inability to complete VOT

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Woolley, BS, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: fMRI phase: 2 fMRI scans - 20IU single administration oxytocin and placebo Chronic Phase: 20IU oxytocin for 3 weeks
- Arm 2: fMRI phase (within subject): 2 fMRI scans - 20IU single administration oxytocin + placebo Chronic Phase: placebo for 3 weeks
- Arm 3: fMRI phase: 2 fMRI scans - 40IU single administration oxytocin + placebo Chronic Phase: 40IU oxytocin for 3 weeks
- Arm 4: fMRI phase: 2 fMRI scans - 40IU single administration oxytocin + placebo Chronic Phase: placebo for 3 weeks
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 7 | 4 | 9 | 6
Completed | 2 | 2 | 6 | 3
Not Completed | 5 | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Only individuals who completed all outcome assessment timepoints were included in the results calculation
Groups:
- Arm 1: fMRI phase: 20IU single administration oxytocin Chronic phase: 20IU oxytocin for 3 weeks
- Arm 2: fMRI phase: 20IU single administration oxytocin Chronic phase: placebo for 3 weeks
- Arm 3: fMRI phase: 40IU single administration oxytocin Chronic phase: 40IU oxytocin for 3 weeks
- Arm 4: fMRI phase: 40IU single administration oxytocin Chronic phase: placebo for 3 weeks
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 2 | 2 | 6 | 3 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 6 | 3 | 13
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 57 [50 to 64] | 60 [55 to 65] | 51 [40 to 64] | 53 [33 to 64] | 54 [33 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 1 | 5
  Male | 2 | 1 | 3 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 4 | 2 | 9
  White | 0 | 1 | 2 | 1 | 4
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 6 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Social Functioning Score
Description: The Social Functioning Scale is a 79-item semi-structured interview based assessment that includes [a global summary score (primary outcome)] The subscale scores of social engagement, interpersonal communication, and prosocial were expected the change in 3 weeks, while other subscales were not expected to change (e.g. employment) and thus were not collected during the chronic period. Scale ranges from 0 to lower functioning to 90 higher functioning.
Time Frame: Baseline visit: Full assessment is collected prior to any treatments fMRI phase: assessment not collected Chronic phase: partial assessment collected before the start (A1) and at end (A2) of 3 weeks of daily administration
Population: Data for an individual was only included if both assessment timepoints were completed in full (i.e. no missing values)
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Arm 2: fMRI phase (within subject): 20IU single administration oxytocin Chronic Phase: placebo for 3 weeks
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 2 | 2 | 6 | 3
score on a scale
  Baseline | 102.5 [98 to 107] | 113.5 [112 to 115] | 79.2 [41 to 97] | 100 [74 to 115]
  A1 | 16 [13 to 19] | 30.5 [30 to 31] | 20.7 [14 to 37] | 20 [19 to 21]
  A2 | 14.5 [13 to 16] | 24 [19 to 29] | 21.3 [12 to 31] | 20 [14 to 30]

2. Secondary Outcome: CAINS Score (Clinical Assessment Interview for Negative Symptoms)
Description: Negative symptoms will be assessed with the CAINS (clinical assessment interview for negative symptoms) comprised of several subscales that will be summed for a global score. Each item is assessed from 0-no impairment to 4-severe deficit. The total score from 0 to 52 where higher scores represent more significant impairment.
Time Frame: Baseline visit: assessment is collected prior to any treatments fMRI phase: assessment not collected Chronic phase: assessment collected before the start (A1) and at end (A2) of 3 weeks of daily administration
Population: Data for an individual was only included if the assessment was completed in full
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 2 | 2 | 5 | 3
score on a scale
  Baseline | 21 [18 to 24] | 6 [5 to 7] | 16.4 [5 to 26] | 20.7 [9 to 41]
  A1 | 19 [14 to 24] | 10.5 [6 to 15] | 18.6 [4 to 31] | 16.7 [8 to 34]
  A2 | 19 [7 to 31] | 10.5 [7 to 14] | 17.2 [1 to 30] | 17 [0 to 36]

3. Other Pre Specified Outcome: QLS Scale (Quality of Life)
Description: Quality of Life will be assessed with the Quality of Life Scale (QLS), a 9-item assessment that measures domains such as interpersonal relations, occupation role functioning, and intrapsychic foundations. Each item is rated from 0 to 6 with the lower values indicating greater severity of symptoms. As such, the total score ranges from 0-54 (higher scores indicate good quality of life).
Time Frame: Baseline visit: assessment not collected fMRI phase: assessment not collected Chronic phase: assessment collected before the start (A1) and at end (A2) of 3 weeks of daily administration
Population: Data for an individual was only included if the assessment was completed in full
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 2 | 2 | 6 | 3
score on a scale
  A1 | 2 [2 to 2] | 6 [4 to 8] | 2.6 [0 to 11] | 4.7 [1 to 10]
  A2 | 2 [1 to 3] | 5.5 [2 to 9] | 3 [0 to 12] | 3 [0 to 7]

4. Other Pre Specified Outcome: Hinting Task
Description: Theory of Mind (ToM) will be assessed using The Hinting Task, a well-validated tool where participants make social inferences after hearing 10 fictional conversations. Each conversation ends with one character's utterance and the participant is asked to determine its meaning.
  Each item is scored from 0 to 2. The summed values of the scale from 0 to 20, where higher values represent better theory of mind / higher functioning
Time Frame: as for outcome 3
Population: Data for an individual was only included if the assessment was completed in full
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 2 | 2 | 6 | 3
score on a scale
  A1 | 19 [19 to 19] | 16 [15 to 17] | 14.8 [0 to 20] | 17.7 [16 to 19]
  A2 | 18.5 [17 to 20] | 16.5 [14 to 19] | 17.4 [8 to 20] | 17.7 [16 to 19]

ADVERSE EVENTS:
Time Frame: approx. 6 weeks: from first visit to final visit
Description: Note: Participants completed 2 phases of the same arm. Including 1 fMRI phase and 1 Chronic Phase. Thus participants are reported twice in this section
Groups:
- Arm 1 fMRI Phase; Arm 2 fMRI Phase: fMRI phase: 20IU single administration oxytocin
- Arm 3 fMRI Phase; Arm 4 fMRI Phase: fMRI phase: 40IU single administration oxytocin
- Arm 1 Chronic Phase: Chronic Phase: 20IU oxytocin for 3 weeks
- Arm 2 Chronic Phase; Arm 4 Chronic Phase: Chronic Phase: placebo for 3 weeks
- Arm 3 Chronic Phase: Chronic Phase: 40IU oxytocin for 3 weeks
Arm/Group | Arm 1 fMRI Phase | Arm 2 fMRI Phase | Arm 3 fMRI Phase | Arm 4 fMRI Phase | Arm 1 Chronic Phase | Arm 2 Chronic Phase | Arm 3 Chronic Phase | Arm 4 Chronic Phase
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/6 | 0/3 | 0/2 | 0/2 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/6 | 0/3 | 0/2 | 0/2 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 1/6 | 0/3 | 0/2 | 0/2 | 1/6 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 fMRI Phase (N=2) | Arm 2 fMRI Phase (N=2) | Arm 3 fMRI Phase (N=6) | Arm 4 fMRI Phase (N=3) | Arm 1 Chronic Phase (N=2) | Arm 2 Chronic Phase (N=2) | Arm 3 Chronic Phase (N=6) | Arm 4 Chronic Phase (N=3)
Pelvic Mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — pt reported a growth near the pelvis and planned to follow up with their regular care team. Growth had been know to the pt prior to receiving study drug, however had not been disclosed during participation

LIMITATIONS AND CAVEATS:
Study did not reach target enrollment numbers needed to achieve target power and statistically reliable results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT03900754/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT03900754/ICF_000.pdf